CLINICAL TRIAL: NCT04026516
Title: Production of a Device to Obtain Continuous Ambulatory Vestibular Assessment (CAVA) - Dizziness Trial
Brief Title: CAVA: Dizziness Trial
Acronym: CAVA
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Staff shortages
Sponsor: Julie Dawson (Other)
Collaborators: University of East Anglia (Other)
Responsible Party: Sponsor-Investigator, Julie Dawson, Research Services Manager, Norfolk and Norwich University Hospitals NHS Foundation Trust
Organization: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 261099 (14-02-19)
Record Dates: First submitted 2019-07-08; First posted 2019-07-19 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Meniere's Disease; Benign Paroxysmal Positional Vertigo; Recurrent Vestibulopathy; Vestibular Migraine
Keywords: eye movements; Electronystagmograpy; nystagmus; electrooculogram; vestibular assessment; ambulatory monitoring
MeSH Terms: conditions — Meniere Disease; Benign Paroxysmal Positional Vertigo; Vestibular Neuronitis; Nystagmus, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAVA Dizziness Trial Arm (Experimental): All trial participants are within this arm. All participants will wear the CAVA device for 30 days and follow the same procedures throughout the trial.
  Interventions: Device: CAVA Device

INTERVENTIONS:
Device: CAVA Device — The CAVA device will be worn continuously for thirty days, during which time it will record eye and head movements

SUMMARY:
Clinical investigation of a medical device (CAVA) for recording eye movements. Patients suffering from diagnosed dizziness conditions will wear the device for 23 hours a day, for 30 days. The device will capture normal eye movement data as well as data corresponding to any dizzy events experienced. At the end of the trial, the data will be downloaded and a scientist will perform a blinded analysis of the data. Specifically, they will attempt to identify the dates on which dizziness was reported.

DETAILED DESCRIPTION:
Dizziness is a common condition that is responsible for a significant degree of material morbidity and burden on our health service. There are multiple causes of dizziness, and these originate from pathologies affecting a large variety of different organ systems. Dizziness is usually episodic and short-lived, so when a patient presents to their health care provider, examination is often normal. As such, diagnosis is challenging and patients often experience significant delay in receiving a diagnosis.

The investigators have developed a prototype device for monitoring dizziness and have tested it in a group of 17 healthy volunteers. The results showed that their device is capable of accurately, precisely and reliably identifying short periods of induced nystagmus (eye movements produced during dizzy attacks) among days' worth of normal eye movement data.

The overall aim of this trial is to test a fully evolved device for the continuous recording of eye movements over a prolonged period of time, on patients suffering from dizziness. For the purpose of this study, the monitoring period is 23 hours a day, for 30 days. The device is composed of two components: a bespoke single-use sensor array that adheres to the participant's face, and a small reusable module that contains a battery, microcomputer, data storage facility, battery and connection port.

The investigators intend to confirm that the device data can be used to identify any occurrence of nystagmus, as produced during attacks of vertigo. Each trial participant will be provided with the device and enough single-use electrode arrays to allow the array to be changed every 24 hours, for thirty days. Participants will be allowed to remove the sensor array for up to 60 minutes each day to allow them to wash and/or shower. If patients experience an episode of dizziness during the trial, they are required to log the details of the event in a trial diary. The identity of these days will not be revealed to the blinded investigator who will later conduct a formal, blinded analysis of the data. At the end of the thirty-day trial, the sensitivity and specificity of the device will be determined by assessing whether the data can be used to correctly identify the dates that participants reported dizziness.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 and over.

* Patients experiencing episodes of true vertigo, with at least two episodes within the preceding month. Relevant medical conditions include Meniere's disease, Benign Paroxysmal Positional Vertigo (BPPV), recurrent vestibulopathy and vestibular migraine.
* Able to commit to 30 days of continuous wear of the trial device as per the study plan.
* Own a telephone.

Exclusion Criteria:

* Potential participants who have a history of dermatological disease, fragile skin, or damage around the forehead.
* Potential participants who have an allergy to plasters and/or medical adhesives - (similarly to materials used in the device).
* History of hypertension or cardiac problems (uncontrolled, acute or de-compensated - phase).
* History of ear disease, or previous ear surgery.
* History of psychotic/neurotic disorders or epilepsy.
* History of eye disease, or previous eye surgery.
* Pregnant or nursing mothers.
* Potential participants who have taken part in a previous CAVA trial.
* Potential participants who are currently taking part in another trial.
* Unable to follow the testing protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Nystagmus detection sensitivity and specificity of 95% | 30 days
  The investigators will determine the sensitivity and specificity of the results obtained by a bespoke computer algorithm for detecting episodes of nystagmus, from data captured by the CAVA device.

SECONDARY OUTCOMES:
Post-trial participant questionnaire | 30 days
  A questionnaire will be provided to the participants at the end of the trial to gather data on device acceptability and other patient feedback. A qualitative assessment of this data will be performed. The device acceptability is measured over 8 questions regarding comfort of wear, ease of wear, self consciousness, effect on sleep with each question having a scale of 1-5. With 5 being the best outcome and 1 being the worst outcome.
Compliance with wearing the device | 30 days
  Investigators will check the participants compliance of wearing the device by using the data in the participants' trial diaries.
Functionality of the device's accelerometer | 30 days
  Data will be downloaded from the device and manually checked to ensure that valid data has been captured.
Functionality of the device's event marker | 30 days
  Data will be downloaded from the device and manually checked to ensure that the known dates and times of event marker activation match the record stored on the device.
Functionality of the device's timestamping capabilities | 30 days
  The known dates and times of event marker activations will be compared to the record stored on the device. From this information, clock drift will be calculated (hh:mm:ss).

CONTACTS AND LOCATIONS:
Overall Officials: John Phillips, Consultant, Principal Investigator — Dr
Locations (1):
- Norfolk & Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom